CLINICAL TRIAL: NCT01193452
Title: A Randomized Phase II Study of Comparing S-1/Leucovorin With sLV5FU2 as the First-line Treatment for Elderly Patients With Colorectal Cancer
Brief Title: S-1/Leucovorin (SL) Versus sLV5FU2 as the First-line Treatment for Elderly Patients With Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Jin Li, Fudan University Shanghai Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-eCRC
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-08

CONDITIONS: Colorectal Cancer
Keywords: elderly patients; advanced colorectal cancer; chemotherapy; S-1; 5-fluorouracil; leucovorin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — S 1 (combination); Leucovorin; Drug Therapy; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-1/LV (Experimental): S-1 combined with Leucovorin
  Interventions: Drug: S-1, Leucovorin
- sLV5FU2 (Active Comparator): 5-FU/LV infusion
  Interventions: Drug: leucovorin, 5-fluorouracil

INTERVENTIONS:
Drug: S-1, Leucovorin — S-1 :
  The initial dosage of S-1 is determined by the body surface area:
  Surface area: 1.25-1.5 m2 : 50mg twice per day;upper than 1.5 m2 : 60mg twice per day
  Leucovorin:
  25mg twice per day po.
  The treatment is given for one week,and no chemotherapy is given for the following one week.
  Other Names: chemotherapy
  Arms: S-1/LV
Drug: leucovorin, 5-fluorouracil — leucovorin: 400mg/m2 intravenous infusion d1;
  5-fluorouracil: 400mg/m2 intravenous push,d1; 2400mg/m2 continuous intravenous infusion for 46 hours
  repeat every 2 weeks
  Other Names: chemotherapy
  Arms: sLV5FU2

SUMMARY:
This phase II trial on the assumption that S-1 combined with Leucovorin may have better efficacy and safety than simplified 5-FU/LV infusion therapy in elderly patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
This is a randomized phase Ⅱ study, in which S-1 is used in combination with leucovorin in elderly patients with advanced colorectal cancer as first-line treatment,comparing with sLV5FU2 therapy. The aim of this study is to determine the efficacy and safety of S-1/LV in elderly patients in the first-line setting. The other secondary endpoints are progression free survival,overall survival, and quality of life are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Oral medication is acceptable
* Histologically confirmed colorectal carcinoma
* Male or female ≥ 65 years of age
* No prior chemotherapy,radiotherapy,target therapy and immunotherapy, except adjuvant chemotherapy with an interval of ≥ 180 days)
* Presence of at least one target lesion measurable by CT scan or MRI,within 15 days prior to trial
* The lab values within 2 weeks prior to trial should meet:

PLT ≥7.5*10^4/mm3 ANC≥2000/mm3 HB≥100g/L Total bilirubin < upper limit of normal level ALT/AST/ALP < 2.5 x UNL (<5 x UNL for patients with liver or bone metastasis) Serum creatinine < UNL

* Performance status (ECOG) 0~1
* Life expectation longer than 90 days

Exclusion Criteria:

* Allergy to S-1,fluorouracil or leucovorin
* Any investigational agent(s) within 4 weeks prior to entry
* Previous or currently exposure to certain drugs which are proved to have influence on blood drug concentration
* Active infection
* Severe organ failures or diseases, including: intestinal obstruction, pulmonary fibrosis, uncontrolled diabetes mellitus,clinically relevant coronary disease, cardiovascular disorder or myocardial infarction,renal or liver failure, severe psychiatric illness,cerebral vascular disease and sever GI ulcer which need blood infusion.
* Uncontrolled hydrothorax,ascites and hydropericardium
* Multiple bone metastatic lesions
* Brain metastases
* Chronic diarrhea or digestive disfunction
* Previous malignancy (except colorectal cancer, history of basal cell carcinoma of skin or pre-invasive carcinoma of the cervix with adequate treatment)
* Strong willingness to receive surgery or highly potential to have intestinal obstruction which may need surgery intervention
* Other conditions that primary investigate or investigator consider to be unsuitable for the trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
response rate | six weeks

SECONDARY OUTCOMES:
progression free survival | six weeks
disease control rate | six weeks
time to treatment failure | six weeks
overall survival | three months
quality of life | six weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD,PhD, Principal Investigator — Fudan University
Locations (1):
- Jin Li', Shanghai, Shanghai Municipality, China